CLINICAL TRIAL: NCT00384293
Title: A Worldwide, Double-Blind, Randomized, Placebo-Controlled Study of MK0524A 2g Coadministered With Intensive LDL-C Lowering Therapy Compared to Intensive LDL-C Lowering Therapy Alone on Carotid Artery Intima Media Thickening (cIMT) in Patients With Heterozygous Familial Hypercholesterolemia (heFH)
Brief Title: Carotid IMT (Intima Media Thickening) Study (0524A-041)(TERMINATED)
Acronym: ACHIEVE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-041; 2006_506
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Results first posted 2009-09-02 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Hypercholesterolemia, Familial
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): MK0524A
  Interventions: Drug: Comparator: niacin (+) laropiprant (MK0524A)
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: Comparator: niacin (+) laropiprant (MK0524A) — niacin (+) laropiprant (2 g) po qd.
  Other Names: MK0524A
  Arms: 1
Drug: Comparator: placebo — niacin (+) laropiprant (2 g) placebo po qd.
  Arms: 2

SUMMARY:
This is a 105-week clinical study in patients with heterozygous familial hypercholesterolemia on intensive Low Density Lipoprotein-cholesterol (LDL-C) lowering therapy intended to assess the affects of MK0524A on carotid intima media thickening using ultrasound compared to patients taking placebo. There will be 12 scheduled clinic visits involving review of medical history, physical exam, vital signs, laboratory testing, ultrasound imaging, and electrocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 to 70 years of age with Heterozygous Familial Hypercholesterolemia and a LDL-C greater than or equal to 100mg/dL and triglycerides less than or equal to 400mg/dL at Visit 1 while on a stable dose of intensive LDL-C lowering therapy

Exclusion Criteria:

* A condition which, in the opinion of the investigator, might pose a risk to the patient or interfere with participating in the study
* Patients with less than 80% drug study compliance
* Patients with chronic medical conditions known to influence serum lipids or lipoproteins or significantly affect the ultrasound acoustic window
* Patients with unstable dose of medications
* Pregnant or lactating women, or women intending to become pregnant are excluded
* Patient with diabetes mellitus that is poorly controlled, or is taking new or recently adjusted antidiabetic pharmacotherapy (with the exception of +/- 10 units of insulin)
* Patients with the following conditions: high grade stenosis (greater than 75%) of the carotid artery, chronic heart failure, uncontrolled/unstable cardiac arrhythmias, unstable hypertension, active or chronic hepatobiliary or hepatic disease, HIV positive, episode of gout (within 1 year)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 937 (Actual)
Dates: Start 2006-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was an MK0524A active run-in period prior to randomization. Per protocol, patients were scheduled to receive MK0524A 1g orally once daily for 4 weeks. The MK0524A dose was then increased to 2g (2x 1g tablets), once daily, for an additional 4 weeks prior to randomization.
Groups:
- MK0524A Active Run-In Period: Patients who received MK0524A during active run-in (Visit 2). Per protocol, patients were scheduled to receive MK0524A 1g orally once daily for 4 weeks. The MK0524A dose was then increased to 2g (2x 1g tablets), once daily, at Visit 3 for an additional 4 weeks prior to randomization.
- MK0524A, 2 g (Postrandomization Period): Patients who were randomized to MK0524A, 2 g (oral administration) once daily.
- Placebo (Postrandomization Period): Patients who were randomized to placebo
Period: MK0524A Active Run-In, Pre-randomization
Arm/Group | MK0524A Active Run-In Period | MK0524A, 2 g (Postrandomization Period) | Placebo (Postrandomization Period)
Started | 937 | 0 | 0
Entered Active run-in, MK0524A 1 g | 937 (Entered active run-in period and received MK0524A 1 g) | 0 | 0
MK0524A Dose Increased to 2 g | 813 (MK0524A dose increased to 2 g in active run-in period) | 0 | 0
Completed | 433 | 0 | 0
Not Completed | 504 | 0 | 0
Not completed — Adverse Event | 120 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 24 | 0 | 0
Not completed — Not cIMT eligible at Visit 3 | 340 | 0 | 0
Not completed — Trial Termination | 16 | 0 | 0
Not completed — Certified Sonographer Not Available | 2 | 0 | 0
Not completed — Patient Unable to Complete cIMT Scan | 1 | 0 | 0
Period: Post-randomization Period
Arm/Group | MK0524A Active Run-In Period | MK0524A, 2 g (Postrandomization Period) | Placebo (Postrandomization Period)
Started | 0 | 214 | 219
Received ≥1 Dose of MK0524A Study Drug | 0 | 214 (Received at least one dose of randomized study drug (All Patients as Treated Population)) | 218
Completed | 0 | 0 | 0
Not Completed | 0 | 214 | 219
Not completed — Adverse Event | 0 | 23 | 7
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 8 | 6
Not completed — Trial Termination | 0 | 180 | 204
Not completed — Patient Randomized in Error | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK0524A, 2 g (Postrandomization Period) | Placebo (Postrandomization Period) | Total
Number analyzed (Participants) | 214 | 218 | 432
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (8.94) | 54.5 (8.22) | 53.8 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 82 | 158
  Male | 138 | 136 | 274

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Carotid Intima Media Thickness
Description: change in mean carotid intima media thickness defined as a composite measure of the left and right common, bulb, and internal carotid artery.
Time Frame: after 96 weeks of postrandomization treatment
Population: study prematurely terminated, no efficacy analyses were performed
Arm/Group | MK0524A Active Run-In Period | MK0524A, 2 g (Postrandomization Period) | Placebo (Postrandomization Period)
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change in Lipid Profile
Time Frame: after 96 weeks of postrandomization treatment
Population: study prematurely terminated, no efficacy analyses were performed
Arm/Group | MK0524A Active Run-In Period | MK0524A, 2 g (Postrandomization Period) | Placebo (Postrandomization Period)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | MK0524A Active Run-In Period | MK0524A, 2 g (Postrandomization Period) | Placebo (Postrandomization Period)
Serious Adverse Events (participants affected / at risk) | 10 | 5 | 8
Other Adverse Events (participants affected / at risk) | 395 | 74 | 54
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | MK0524A Active Run-In Period | MK0524A, 2 g (Postrandomization Period) | Placebo (Postrandomization Period)
Acute coronary syndrome (Cardiac disorders) | 0/937 | 0/214 | 1/218
Acute myocardial infarction (Cardiac disorders) | 1/937 | 0/214 | 0/218
Acute pectoris (Cardiac disorders) | 0/937 | 1/214 | 0/218
Angina unstable (Cardiac disorders) | 1/937 | 1/214 | 1/218
Atrial fibrillation (Cardiac disorders) | 1/937 | 0/214 | 0/218
Myocardial infarction (Cardiac disorders) | 1/937 | 0/214 | 0/218
Pancreatitis (Gastrointestinal disorders) | 0/937 | 0/214 | 1/218
Constipation (Gastrointestinal disorders) | 1/937 | 0/214 | 0/218
Pyrexia (General disorders) | 0/937 | 0/214 | 1/218
Hepatitis (Hepatobiliary disorders) | 1/937 | 0/214 | 0/218
Anaphylactic shock (Immune system disorders) | 0/937 | 0/214 | 1/218
Diverticulitis (Infections and infestations) | 1/937 | 0/214 | 0/218
Staphylococcal sepsis (Infections and infestations) | 1/937 | 0/214 | 0/218
Limb injury (Injury, poisoning and procedural complications) | 0/937 | 0/214 | 1/218
Hypoglycaemia (Metabolism and nutrition disorders) | 1/937 | 0/214 | 0/218
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0/937 | 2/214 | 0/218
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0/937 | 1/214 | 1/218
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/937 | 0/214 | 1/218
Toe deformity (Musculoskeletal and connective tissue disorders) | 0/937 | 0/214 | 1/218
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/937 | 0/214 | 0/218
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/937 | 0/214 | 0/218
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/937 | 0/214 | 1/218
Renal failure acute (Renal and urinary disorders) | 1/937 | 0/214 | 0/218
Ovarian cyst (Reproductive system and breast disorders) | 0/937 | 1/214 | 0/218
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/937 | 0/214 | 1/218
Arterial stenosis (Vascular disorders) | 1/937 | 0/214 | 0/218
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | MK0524A Active Run-In Period | MK0524A, 2 g (Postrandomization Period) | Placebo (Postrandomization Period)
Diarrhoea (Gastrointestinal disorders) | 20/937 | 8/214 | 4/218
Nausea (Gastrointestinal disorders) | 24/937 | 5/214 | 0/218
Vomiting (Gastrointestinal disorders) | 0/937 | 5/214 | 0/218
Fatigue (General disorders) | 0/937 | 6/214 | 5/218
Influenza (Infections and infestations) | 0/937 | 14/214 | 18/218
Nasopharyngitis (Infections and infestations) | 23/937 | 14/214 | 13/218
Upper respiratory tract infection (Infections and infestations) | 0/937 | 4/214 | 6/218
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/937 | 8/214 | 3/218
Back pain (Musculoskeletal and connective tissue disorders) | 0/937 | 8/214 | 6/218
Myalgia (Musculoskeletal and connective tissue disorders) | 0/937 | 6/214 | 8/218
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/937 | 2/214 | 7/218
Headache (Nervous system disorders) | 52/937 | 10/214 | 5/218
Paraesthesia (Nervous system disorders) | 47/937 | 0/214 | 0/218
Burning Sensation (Nervous system disorders) | 25/937 | 0/214 | 0/218
Dizziness (Nervous system disorders) | 21/937 | 0/214 | 0/218
Pruritus (Skin and subcutaneous tissue disorders) | 78/937 | 10/214 | 2/218
Erythema (Skin and subcutaneous tissue disorders) | 23/937 | 0/214 | 0/218
Rash (Skin and subcutaneous tissue disorders) | 22/937 | 0/214 | 0/218
Flushing (Vascular disorders) | 184/937 | 5/214 | 0/218
Hot flush (Vascular disorders) | 37/937 | 0/214 | 0/218

LIMITATIONS AND CAVEATS:
After a detailed review of pooled carotid IMT data from contemporary studies, the Steering Committee recommended that Merck prematurely stop the study; as designed, the study was significantly underpowered. Efficacy analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.